CLINICAL TRIAL: NCT03338231
Title: Clinical Study of Immunity Duration of Yellow Fever Vaccine in Military, Participants of "Dose-response Study of Yellow Fever Vaccine 17DD Produced by Bio-Manguinhos / Fiocruz" in 2009
Brief Title: Clinical Study of Immunity Duration of Yellow Fever Vaccine in Military
Status: Completed | Type: Observational
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Other Study IDs: ASCLIN 001/2017
Record Dates: First submitted 2017-11-01; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Yellow Fever Vaccine
Keywords: Immunity duration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Yellow fever is an acute viral disease transmitted by mosquitoes in South America, Central America and Africa. It is more prevalente in males gender and the age above 15 years due to the greater exposure in the wild endemic area of yellow fever.

According to the World Health Organization (WHO), a single dose of the yellow fever vaccine is sufficient to maintain protective immunity against yellow fever for a lifetime, therefore a booster dose is not required. This issue is difficult to evaluate because there is no serological correlate of protection against yellow fever and seropositivity is defined with several cut-off points. Although studies indicate that the duration of protection after vaccination is long, many studies have demonstrated a reduction of the antibody titrer over the years. Consequently, there is more concern about people who live in endemic areas. For this reason, Brazil recommends revaccinating once at least until additional studies are performed.

It is important to know the duration of immunity induced by lower doses of YF vaccine. In our knowledge, there is a lack of clinical studies evaluating the immunity duration of the yellow fever vaccine with lower doses. This information is relevant to subsidize the routine recommendation of YF vaccine fractional dose for adults.

DETAILED DESCRIPTION:
This is an observational study in young adult males who received the first dose of the yellow fever vaccine in 2009 when they participated in the "Dose-response study of the yellow fever vaccine 17DD produced by Bio-Manguinhos / Fiocruz.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the "Dose-response study of the yellow fever vaccine 17DD produced by Bio-Manguinhos / Fiocruz" in 2009.
* Not been revaccinated during the "Dose-response study of the yellow fever vaccine 17DD produced by Bio-Manguinhos / Fiocruz" of 2009.
* Not having received another dose of the 17DD yellow fever vaccine after participating in the 2009 "Bio-Manguinhos / Fiocruz" 17DD yellow fever vaccine dose-response study.
* Provide name, address, telephone and other information so that you can contact if necessary.
* Ability to understand and sign the TCLE.

Exclusion Criteria:

* Impossibility or refusal to collect blood

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Male adults who received the first dose of the yellow fever vaccine in 2009 when they participated in the "Dose-response study of the yellow fever vaccine 17DD produced by Bio-Manguinhos / Fiocruz
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Number of seropositivity participants to YF vaccine as assessed by PRNT. | 8 years after the 1 st dose of yellow fever vaccine
  To evaluate the seropositivity by the means of the neutralizing antibody dosage in the participants of the "Dose-response study of the 17DD yellow fever vaccine produced by Bio-Manguinhos/Fiocruz" realized in 2009

SECONDARY OUTCOMES:
Individual repertoire of immunoglobulins profile as assessed by the PEPperPRINT and phenotypic/functional anti-amaryl memory cell analyse. | 8 years after the 1 st dose of yellow fever vaccine
  To evaluate individual repertoire of immunoglobulins profile directed to amaryl epitopes by the PEPperPRINT (PEPperCHIP® Yellow Fever Virus Proteome Microarrays) Guidelines and to evaluate the phenotypic and funcional profile of anti-yellow memory cell in the participants of the "Dose-response study of the 17DD yellow fever vaccine produced by Bio-Manguinhos/Fiocruz" realized in 2009

CONTACTS AND LOCATIONS:
Overall Officials: Reinaldo M Martins, PhD, Principal Investigator — Oswaldo Cruz Foundation
Locations (1):
- Bio-Manguinhos/Fiocruz, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Menezes Martins R, Maia MLS, de Lima SMB, de Noronha TG, Xavier JR, Camacho LAB, de Albuquerque EM, Farias RHG, da Matta de Castro T, Homma A; Collaborative Group for Studies on Duration of Immunity from Yellow Fever Vaccine. Duration of post-vaccination immunity to yellow fever in volunteers eight years after a dose-response study. Vaccine. 2018 Jun 27;36(28):4112-4117. doi: 10.1016/j.vaccine.2018.05.041. Epub 2018 May 18. PMID 29784469